CLINICAL TRIAL: NCT06382688
Title: The Effects of IV Administration of ChromaDex's Niagen®, Nicotinamide Riboside Chloride as Compared to IV Administration of NAD+: A Randomized, Placebo Controlled Clinical Trial
Brief Title: IV Administration of ChromaDex's Niagen® as Compared to NAD+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23-08-0010
Record Dates: First submitted 2024-04-04; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy Aging
Keywords: nicotinamide adenine dinucleotide; nicotinamide riboside chloride; Niagen
MeSH Terms: interventions — NAD; nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NR (Cohorts 1&2) (Experimental): IV administered 500 mg of sterile Niagen® (nicotinamide riboside chloride) diluted, in 500 ml of saline
  Interventions: Dietary Supplement: Niagen® (nicotinamide riboside) IV
- Active Comparator (Cohorts 1&2) (Active Comparator): IV administered 500 mg of sterile nicotinamide adenine dinucleotide in 500 ml of saline
  Interventions: Dietary Supplement: NAD+ (nicotinamide adenine dinucleotide) IV
- Oral Comparator (Cohort 1 only) (Other): orally administered 500 mg of sterile Niagen® (nicotinamide riboside chloride) in capsules
  Interventions: Dietary Supplement: Niagen® (nicotinamide riboside) oral
- Placebo (Cohort 1 only) (Placebo Comparator): IV administered 500 ml of saline
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: NAD+ (nicotinamide adenine dinucleotide) IV — NAD+ enables cells to generate cellular energy from the food that one eats
  Other Names: NAD+
  Arms: Active Comparator (Cohorts 1&2)
Dietary Supplement: Niagen® (nicotinamide riboside) IV — NR is a unique member of the vitamin B3 family. Cells can use NR to create nicotinamide adenine dinucleotide (NAD+), which is an essential molecule found in every living cell. Patients in this arm received an IV administration.
  Arms: NR (Cohorts 1&2)
Dietary Supplement: Niagen® (nicotinamide riboside) oral — NR is a unique member of the vitamin B3 family. Cells can use NR to create nicotinamide adenine dinucleotide (NAD+), which is an essential molecule found in every living cell. Patients in this arm received an oral administration.
  Other Names: Niagen® (oral)
  Arms: Oral Comparator (Cohort 1 only)
Other: Placebo — These individuals received a saline IV
  Arms: Placebo (Cohort 1 only)

SUMMARY:
This is a 2-part study evaluating the effects of IV administration of NR on healthy adult populations. Study 1 involved all four arms with 37 people. The second study only included the active NR and NAD+ arms to further evaluate tolerability and comfort of the IV.

DETAILED DESCRIPTION:
The purpose of this work is to establish and quantify the safety and efficacy of IV administration of ChromaDex's Niagen®, nicotinamide riboside chloride in comparison to currently available IV NAD+, a saline IV, and orally administered Niagen®

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness and demonstrated ability to comply with all study procedures, as well as availability for the duration of the study
* Lives within 100 miles of a NRI study site
* Any gender, aged 40+ (For the 5th arm, only males will be evaluated.)
* Good general health as evidenced by medical history
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional month after the end of the study
* Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

* Current diagnosis of any seizure disorder, diabetes or insulin resistance, any kidney or liver disorder, heart disease, cancer, or Parkinson's disease,
* Pregnancy, trying to conceive, or breastfeeding
* Known allergic reactions to any components of the intervention
* Positive COVID-19 test within 30 days of the study period
* Recent dramatic weight changes (10% change in body weight in the last 6 months)
* Existing usage of a NAD+ or NAD precursor supplement in any form.
* Introducing a new investigational drug or other intervention within 30 days before the start of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | immediately before the intervention, immediately after the intervention, 3 and 6 hours post-intervention, and at the 24 hour visit.
  blood pressure, systolic and diastolic, will be measured
Heart rate | immediately before the intervention, immediately after the intervention, 3 and 6 hours post-intervention, and at the 24 hour visit.
  heart rate will be measured
Total NAD measured through dried blood spot testing | Blood spot data is collected at baseline, immediately after the intervention, 3 hours after the intervention, 6 hours after the intervention,on day 2, 7, and 14.
  NAD analysis will be developed from dried blood spots obtained by pricking a finger
Glucose | baseline, at 3 hours, and 24 hours post administration of intervention
  Total glucose in blood via mg/dL
Insulin Levels | baseline, at 3 hours, and 24 hours post administration of intervention
  Total insulin in blood via mcU/mL
total NAD measured through blood and plasma | baseline, at 3 hours, and 24 hours post administration of intervention
  NAD analysis conducted on whole blood and plasma samples
Tolerable Infusion Rate | through intervention completion, an average of 2 hours
  The total amount of time it takes patients to comfortably receive the IV

SECONDARY OUTCOMES:
Complete Blood Count | baseline, at 3 hours, and 24 hours post administration of intervention
  A complete blood count with differential will be evaluated through whole blood samples
Comprehensive Metabolic Panel | baseline, at 3 hours, and 24 hours post administration of intervention
  comprehensive metabolic panel will be evaluated through whole blood samples
Sleep Scale | Change from baseline at day 14
  This is a validated scale measuring 7 subdomains of sleep. It is measured on a likert scale. Scores on each subdomain can range from 5-42 with higher scores indicating greater quality of sleep
Energy Scale | Change from baseline at day 14
  This is a validated scale measuring 6 subdomains of energy. It is measured on a likert scale. Scores on each subdomain can range from 5 to 42, with higher scores indicating greater energy levels.

OTHER OUTCOMES:
Subjective Experience | Immediately after the intervention, 24 hours after the intervention, 7 days after the intervention, and 14 days after the intervention
  Patients will be asked open ended questions to describe the experience of receiving the IV or oral intake of the assigned product.

CONTACTS AND LOCATIONS:
Locations (1):
- Nutraceuticals Research Institute, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Patient consent does not include data sharing outside of pre-specified organizations.